CLINICAL TRIAL: NCT07373041
Title: Implementation Testing of the Heart Failure Carer Support Programme in the United Kingdom.
Brief Title: Heart Failure Carer Support Programme: Implementation Testing in the UK.
Acronym: HELP
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Queen's University, Belfast (Other)
Collaborators: Belfast Health and Social Care Trust (Other); Southern Health and Social Care Trust (Other Government); South Eastern Health and Social Care Trust (Other); King's College Hospital NHS Trust (Other); Glasgow Royal Infirmary (Other)
Responsible Party: Principal Investigator, Gareth Thomson, Project Manager, Queen's University, Belfast
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: B25/04
Record Dates: First submitted 2026-01-07; First posted 2026-01-28 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Heart Failure; Care Givers; Self Management
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Carers (Experimental): 180 informal carers of people with symptomatic heart failure across the three collaborating centres (Northern Ireland, England, and Scotland). These carers will receive the HEart faiLure carer support Programme (HELP).
  Interventions: Behavioral: HEart faiLure carer support Programme (HELP)
- Patients with symptomatic heart failure (No Intervention): The patients who are receiving support from the recruited carers will be invited to provide outcome data (approximately 180), which will enable an assessment of the dyadic impact of HELP.

INTERVENTIONS:
Behavioral: HEart faiLure carer support Programme (HELP) — A 6-week, psychoeducational intervention consisting of two components: 1) Online support group sessions and 2) Educational booklet and supplementary website. A weekly online support group session will be delivered over 6 weeks via ZOOM by local specialist heart failure nurses. Each session will consist of 12 carers and last approximately 60 minutes. The sessions will initiate with a presentation (approximately 20 minutes in duration) on the allocated topic, including questions and group discussions throughout.
  Carers will complete self-directed learning across the educational booklet and website, which will complement the support group sessions.
  Arms: Carers

SUMMARY:
Background:

Heart failure (HF) is widespread in the United Kingdom (UK). Many of these patients rely on support from family carers who are ill-prepared and supported for this role. These carers often experience poor mental and physical health because of their caring role. HEart faiLure carer support Programme (HELP) is the first intervention in the UK developed with carers of patients with HF to support them with looking after themselves and the patients they care for.

Aim:

To identify the best way of delivering HELP to all carers across the UK and evaluate its impact on carers and patients.

Methods:

HF Nurses will deliver HELP across 3 sites in the UK to approximately 180 carers of patients with HF. The carers targeted will be those who require additional support (caring for a patient who has HF symptoms). These carers will be nominated for the project by patients identified by nurses at in- and out-patient HF appointments. These patients (around 180) will also be invited to provide information for the project. HELP includes 6 online educational support sessions (1 hour each) delivered weekly, along with an educational booklet and website that provide additional support and advice. We will evaluate the impact of HELP on outcomes for patients (i.e., hospital admissions, GP visits, and quality of life) and carers (i.e., burden, preparedness, and quality of life). Interviews and logs / questionnaires will be completed by participants and staff, which will help us understand how best to deliver HELP. Information for the project will be collected at baseline, during HELP, immediately post-HELP (6 weeks), and 6 months after finishing HELP.

Impact:

The findings will allow us to develop a plan for giving HELP to all carers throughout the UK to provide them with the education and support they need.

ELIGIBILITY:
Carers

Inclusion Criteria

1. Aged 18 years or older
2. Physical and mental ability to operate a digital device, engage comfortably in conversation with peers, and be able to read written materials
3. Caring (regular, unpaid care) for a person with a clinical diagnosis of heart failure (HF) who is receiving standard evidence-based HF therapies and has either HF symptoms or 1 episode of decompensation (symptoms requiring medical attention) in previous 6 months
4. Ability to speak and understand English

Exclusion criteria

1. Lacking capacity to give consent
2. Under the age of 18

Patients

Inclusion Criteria

1. Aged 18 years or older
2. Physical and mental ability to engage comfortably in conversation and be able to read written materials
3. Clinical diagnosis of HF and receiving standard evidence-based HF therapies and has either HF symptoms or 1 episode of decompensation (symptoms requiring medical attention) in previous 6 months
4. Ability to speak and understand English
5. Receiving regular, unpaid support with managing his / her condition from a loved one or friend (e.g., a relative or spouse)

Exclusion criteria

1. Lacking capacity to give consent
2. Under the age of 18
3. Carer refused to participate in HELP

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 360 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2027-08-01 (Estimated); Study Completion 2027-09-01 (Estimated)

PRIMARY OUTCOMES:
Participant-reported experiences of fidelity of HELP implementation assessed by semi-structured interviews following a study-specific topic guide. | 6 months
  Semi-structured, audio-recorded interviews will be conducted with participants (carers, patients, and healthcare professionals). The study-specific interview guide will include open-ended questions exploring: 1) Study Design, 2) Provider Training, 3) Intervention Delivery, 4) Treatment Receipt, and 5) Enactment. Interviews will be conducted via a telephone call (approximately 45-60 minutes in duration). Interviews will be transcribed verbatim and analysed with adaptive framework analysis.
Participant-reported experiences of contextual factors influencing HELP implementation assessed by semi-structured interviews following a study-specific topic guide. | 6 months
  Semi-structured, audio-recorded interviews will be conducted with participants (carers, patients, and healthcare professionals). The study-specific interview guide will include open-ended questions exploring barriers and facilitators to HELP implementation. Interviews will be conducted via a telephone call (approximately 45-60 minutes in duration). Interviews will be transcribed verbatim and analysed with adaptive framework analysis.
Cost of HELP implementation. | Baseline to 1 year
  The economic cost of HELP implementation in the UK will be estimated via the collection of data detailing training costs and time input for supervision of HELP facilitators, along with Facilitator logs each session documenting time, expenditure, resources required, and adaptations made for individual carers.

SECONDARY OUTCOMES:
Change in score from baseline in Zarit Burden Interview, Short Form | Baseline, 6 weeks, and 6 months
  Completed by carers.
Change in score from baseline in Preparedness for Caregiving Scale | Baseline, 6 weeks, and 6 months
  Completed by carers
Change in score from baseline in 12-Item Short Form Survey | Baseline, 6 weeks, and 6 months
  Completed by carers
Change in score from baseline in Hospital Anxiety and Depression Scale | Baseline, 6 weeks, and 6 months
  Completed by carers
Change in score from baseline in Perceived Stress Scale | Baseline, 6 weeks, and 6 months
  Completed by carers
Change in score from baseline in Multidimensional Scale of Perceived Social Support | Baseline, 6 weeks, and 6 months
  Completed by carers
Change in score from baseline in Minnesota Living with Heart Failure Questionnaire | Baseline, 6 weeks, and 6 months
  Completed by patients
Change in score from baseline in EuroQol Five Dimension Questionnaire | Baseline, 6 weeks, and 6 months
  Completed by patients
Number of hospital admissions and GP visits with reasons over previous 6 months | Baseline and 6 months
  For patients
Perspectives on how HELP has influenced behaviour | Week 1, week 2, week 3, week 4, week 5, and week 6
  Data collected via bespoke questionnaires completed by carers and patients
Perspectives on long-term adherence to support provided by HELP | 6 months
  Collected via a questionnaire completed by carers and patients

IPD SHARING:
Plan to Share IPD: Yes
Consent will be obtained from participants for data preservation and sharing in an anonymised format. As per the QUB Research Data Management Policy [https://www.qub.ac.uk/directorates/InformationServices/TheLibrary/CustomerService/PoliciesandRegulations/ResearchDataManagementPolicy/], data will be retained in an anonymised format for a minimum of 5 years following publication if they are of continuing value to the researchers and the wider research community. Upon project completion, data sets will be allocated a DOI and transferred to QUB's research information management system (Pure) for long-term preservation, which will contain links to the project and relevant publications. All data that may identify participants will be destroyed following QUB procedures. Data will be exclusive to the team until project completion. After which, data may be shared in an anonymised format with participant consent.
Supporting Information: Study Protocol
Time Frame: With participant consent, data sets will be shared following project completion (approximately December 2027). These data sets will be retained by QUB indefinitely.
Access Criteria: Data will be exclusive to the team until project completion. After which, any data collected may be shared in an anonymised format with participant consent.
URL: https://www.qub.ac.uk/directorates/InformationServices/TheLibrary/CustomerService/PoliciesandRegulations/ResearchDataManagementPolicy/